CLINICAL TRIAL: NCT00381199
Title: Nabilone Versus Amitriptyline in Improving Quality of Sleep in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GEN#05-017
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Fibromyalgia; Sleep Initiation and Maintenance Disorders
Keywords: fibromyalgia; cannabinoid; chronic pain; sleep; insomnia; diffuse widespread pain; antidepressant
MeSH Terms: conditions — Fibromyalgia; Sleep Initiation and Maintenance Disorders; Chronic Pain | interventions — Amitriptyline; nabilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Amitriptyline Hydrochloride
Drug: Nabilone

SUMMARY:
Most chronic pain patients with insomnia are currently not well-managed using existing medications. If found to safely improve sleep with chronic pain patients, nabilone could be added to the treatment options available in the management of fibromyalgia and associated symptoms.

The principle hypothesis of this study is that nabilone at a dose of 0.5-1mg is as efficacious as amitriptyline at a dose of 10-20mg, in improving sleep quality in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years;
* A diagnosis of fibromyalgia according to the American College of Rheumatology classification criteria (Wolfe F, Smythe HA, et al 1990);
* Suffering from self-reported disturbed sleep;
* Negative urine screen for cannabinoids;
* Women of childbearing potential must agree to use adequate contraception during study and for 3 months after study;
* Ability to attend research centre every second week for approximately seven to nine weeks and be able to be contacted by telephone during the study period;
* Stable drug regimen for 1 month prior to randomization;
* Normal liver (AST <3x normal) and renal function (serum creatinine <133µmol/L);
* Haematocrit >38%;
* Negative serum bHCG;
* Proficient in English or French;
* Willing and able to give written informed consent;
* Ability to follow study protocol (cognitive and situational).

Exclusion Criteria:

* Patients currently using cannabis or cannabinoid or tricyclic antidepressants (TCA) and who are unable to undergo a 2 week washout period before entering the study;
* Pain due to cancer;
* Unstable cardiac disease such as cardiac arrhythmias, cardiac failure, ischaemic heart disease and/or hypertension on clinical history and examination;
* History of psychotic disorder or schizophrenia;
* Known hypersensitivity to cannabinoids, amitriptyline, or related tricyclic antidepressants;
* Currently taking or unable to stop taking monoamine oxidase inhibitors (a two-week washout period is necessary for subjects taking MAOIs);
* History of seizures/epilepsy;
* Diagnosis of glaucoma;
* Urinary retention;
* Pregnancy and/or breast-feeding;
* Participation in other clinical trial in the 30 days prior to randomization;
* A recent manic episode (within the past year);
* Current suicidal ideation or history of suicide attempts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Quality of sleep assessed using the Leeds Sleep Evaluation Questionnaire and the Insomnia Severity Index | Day 1, 15, 29 and 43 and given to the patient to complete every second day while taking the study medication

SECONDARY OUTCOMES:
Pain Intensity using the VAS (visual analogue scale) | Days 1, 15, 29 and 43
Pain Quality using the McGill Pain Questionnaire | Days 1, 15, 29 and 43
Mood using the Profile of Mood States (POMS) Questionnaire | Days 1, 15, 29 and 43
Quality of Life using the Fibromyalgia Impact Questionnaire (FIQ) | Days 1, 15, 29 and 43

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Ware, Principal Investigator — McGill University Health Centre, Pain Centre
Locations (1):
- McGill University Health Centre, Pain Centre, Montreal, Quebec, Canada